CLINICAL TRIAL: NCT02537470
Title: A 12-week Randomized, Double-blind, Parallel-group, Placebo-controlled Study to Determine the Efficacy and Safety of Biphasic Remogliflozin Etabonate When Administered to Subjects With Type 2 Diabetes Mellitus
Brief Title: Safety and Efficacy of Biphasic Remogliflozin Etabonate in the Treatment of Type 2 Diabetes
Acronym: BRID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BHV Pharma (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV20200
Record Dates: First submitted 2015-08-25; First posted 2015-09-01 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Other): Placebo
  Interventions: Other: Placebo
- Arm 2 (Experimental): Biphasic remogliflozin etabonate
  Interventions: Drug: Biphasic Remogliflozin Etabonate

INTERVENTIONS:
Drug: Biphasic Remogliflozin Etabonate — Experimental Drug
  Arms: Arm 2
Other: Placebo — Placebo Comparator
  Arms: Arm 1

SUMMARY:
This is a dose-ranging study to evaluate the efficacy, safety and tolerability of a range of doses of a biphasic formulation of remogliflozin etabonate compared to placebo, administered over 12 weeks in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Subject with clinical diagnosis of type 2 diabetes
* HbA1c 7.0 - 10.5% inclusive at Visit 1.

Exclusion Criteria:

* History of metabolic acidosis or ketoacidosis.
* Current active renal disease that is not related to hypertension or type 2 diabetes (e.g. non-diabetic glomerulonephritis, interstitial nephritis, symptomatic nephrolithiasis, etc.)
* Use of an investigational device or investigational drug within 30 days or 5 half-lives (whichever is longer) prior to Visit 1.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2015-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Glycosylated haemoglobin A1c (HbA1c) at Week 12 | 12 weeks

SECONDARY OUTCOMES:
HbA1c | at weeks 4, 8 and 12
Fasting plasma glucose (FPG) | at Weeks 4, 8 and 12
Insulin | at Weeks 4, 8 and 12
C-peptide | at Weeks 4, 8 and 12
Total Cholesterol | at Weeks 4, 8 and 12
LDL-c | at Weeks 4, 8 and 12
HDL-c | at Weeks 4, 8 and 12
Serum Triglycerides | at Weeks 4, 8 and 12
Body Weight | at Weeks 4, 8 and 12
Waist Circumference | at Weeks 4, 8 and 12
Adverse Events (AE) | Over 12 weeks
Safety endpoints include AEs, incidence of urinary tract infections, incidence of genital fungal infections, vital signs, ECGs and standard laboratory tests | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Neutel, MD, Principal Investigator — Orange County Research Center
Locations (19):
- United States (19):
  - Advanced Arizona Clinical Research, Tucson, Arizona
  - Long Beach Clinical Trials, Long Beach, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - National Research Institute, Los Angeles, California
  - Orange County Research Center, Tustin, California
  - Diablo Clinical Research, Walnut Creek, California
  - Chase Medical Research, Waterbury, Connecticut
  - Medical Research Unlimited, Hialeah, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Meridien Research, Tampa, Florida
  - eStudySite, Las Vegas, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Albuquerque Clinical Trials, Inc, Albuquerque, New Mexico
  - Mountain View Clinical Research, Greer, South Carolina
  - New Phase Research & Development, Knoxville, Tennessee
  - Austin Center for Clinical Research, Austin, Texas
  - Padre Coast Clinical Research, Corpus Christi, Texas
  - Juno Research, LLC, Houston, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah